CLINICAL TRIAL: NCT03887520
Title: Multi-center Cross-sectional Epidemiological Study to Characterize the Prevalence and Distribution of Lipoprotein(a) Levels Among Patients With Established Cardiovascular Disease
Brief Title: Lipoprotein(a) in Patients With Cardiovascular Disease (CVD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTQJ230A12001; 2018-003786-34 (EudraCT Number)
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Disease and Lipoprotein(a)
Keywords: CVD, Lipoprotein (a),
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a multi-center cross-sectional epidemiological study to estimate the prevalence (%) of patients with elevated Lp(a) in patients with established CVD defined by their medical history. One study visit is planned for data collection. Relevant medical history and laboratory values for LDL-cholesterol (LDL-C) and Lp(a) within a past pre-specified period will be collected retrospectively. In case laboratory data are not available, blood sampling will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiovascular disease (Other): Patients with established Cardiovascular disease
  Interventions: Diagnostic Test: Blood draw for Lp(a)

INTERVENTIONS:
Diagnostic Test: Blood draw for Lp(a) — Collect sample for Lipoprotein(a) testing
  Other Names: In case retrospective laboratory data are not available, blood sampling will be performed to analyze Lp(a)

SUMMARY:
The study is conducted to improve knowledge about the epidemiology of Lipoprotein(a) in patients with established cardiovascular disease (CVD).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Established CVD defined as one of the following:

  * History of a myocardial infarction (MI) ≥3 months and ≤10 years before the study visit
  * History of ischemic stroke ≥ 3 months and ≤ 10 years before the study visit
  * Symptomatic PAD (intermitted claudication with ankle-brachial index ≤0.90 and/or lower limb amputation or re-vascularization due to lower limb ischemia

Exclusion Criteria:

- Patients currently enrolled in clinical studies with investigational drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49001 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with normal and elevated Lipoprotein(a) (Lp(a)) levels in patients with established Cardiovascular Disease (CVD) | At screening
  Prevalence of normal and elevated Lp(a) levels in patients with established CVD

SECONDARY OUTCOMES:
Lipoprotein(a) (Lp(a)) values | At screening
  Evaluate the median and other relevant statistics describing the distribution of Lp(a) within the normal range and elevated Lp(a) levels
Lp(a) values by region and country | At screening
  Evaluate the median and other relevant statistics describing the distribution of Lp(a) by region and country
Low-density lipoprotein cholesterol (LDL(C)) values (corrected and uncorrected) | At screening
  Evaluate the median and other relevant statistics describing the distribution of LDL-C (corrected and uncorrected) within the normal range and with elevated Lp(a) levels

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (723):
- United States (153):
  - Novartis Investigative Site, Andalusia, Alabama
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Cottonwood, Arizona
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Surprise, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Concord, California
  - Novartis Investigative Site, Covina, California
  - Novartis Investigative Site, Fresno, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Orangevale, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, West Hills, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Bridgeport, Connecticut
  - Novartis Investigative Site, Hartford, Connecticut
  - Novartis Investigative Site, Waterbury, Connecticut
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Brandon, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Saint Augustine, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Dunwoody, Georgia
  - Novartis Investigative Site, Thomasville, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Lombard, Illinois
  - Novartis Investigative Site, Park Ridge, Illinois
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Iowa City, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Hammond, Louisiana
  - Novartis Investigative Site, Houma, Louisiana
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Zachary, Louisiana
  - Novartis Investigative Site, Scarborough, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Ft. Washington, Maryland
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Bingham Farms, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Flint, Michigan
  - Novartis Investigative Site, Grand Blanc, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Midland, Michigan
  - Novartis Investigative Site, Petoskey, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Wyoming, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Belzoni, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Southaven, Mississippi
  - Novartis Investigative Site, Yazoo City, Mississippi
  - Novartis Investigative Site, City of Saint Peters, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Lebanon, New Hampshire
  - Novartis Investigative Site, Nashua, New Hampshire
  - Novartis Investigative Site, Ridgewood, New Jersey
  - Novartis Investigative Site, Summit, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Binghamton, New York
  - Novartis Investigative Site, Endwell, New York
  - Novartis Investigative Site, Manhasset, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, North Massapequa, New York
  - Novartis Investigative Site, Riverhead, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Morehead City, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Sanford, North Carolina
  - Novartis Investigative Site, Shelby, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Lancaster, Pennsylvania
  - Novartis Investigative Site, Lansdale, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Yardley, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Novartis Investigative Site, Summerville, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, Marshall, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Sugar Land, Texas
  - Novartis Investigative Site, Temple, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Novartis Investigative Site, Layton, Utah
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Manassas, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Argentina (15):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Caba
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, Santa Fe
- Australia (6):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Perth, Western Australia
- Austria (5):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (8):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Dendermonde
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Mechelen
  - Novartis Investigative Site, Tienen
- Brazil (21):
  - Novartis Investigative Site, Maceió, Alagoas
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Maringá, Paraná
  - Novartis Investigative Site, Caxias do Sul, Porto Alegre
  - Novartis Investigative Site, Canoas, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Aracaju, Sergipe
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Bulgaria (11):
  - Novartis Investigative Site, Blagoevgrad
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Kardzhali
  - Novartis Investigative Site, Pazardzhik
  - Novartis Investigative Site, Pernik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (19):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Oakville, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Chicoutimi, Quebec
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Québec
- Chile (3):
  - Novartis Investigative Site, Viña del Mar, Región de Valparaíso
  - Novartis Investigative Site, Santiago, RM
  - Novartis Investigative Site, Santiago
- China (14):
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (9):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Medellín
  - Novartis Investigative Site, Pasto
  - Novartis Investigative Site, San Gil
- Czechia (31):
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Český Krumlov, Czech Republic
  - Novartis Investigative Site, Jablonec nad Nisou, Czech Republic
  - Novartis Investigative Site, Kroměříž, Czech Republic
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Pardubice, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Znojmo, Czech Republic
  - Novartis Investigative Site, Most, CZE
  - Novartis Investigative Site, Trutnov, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Broumov
  - Novartis Investigative Site, CZE
  - Novartis Investigative Site, Hlučín
  - Novartis Investigative Site, Hodonín
  - Novartis Investigative Site, Jihlava
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Ostrava
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Přerov
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Valašské Meziříčí
- Denmark (6):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Arhus N
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Viborg
- Egypt (3):
  - Novartis Investigative Site, Aswān, EGY
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
- France (20):
  - Novartis Investigative Site, Auxerre
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Compiègne
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Le Coudray
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valenciennes
- Germany (58):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gelnhausen
  - Novartis Investigative Site, Goch
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Koeln-Nippes
  - Novartis Investigative Site, Künzing
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Meißen
  - Novartis Investigative Site, Memmingen
  - Novartis Investigative Site, Muehldorf Am Inn
  - Novartis Investigative Site, Mühldorf
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Northeim
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Saint Ingbert - Oberwuerzbach
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wangen
  - Novartis Investigative Site, Warendorf
  - Novartis Investigative Site, Wedel
  - Novartis Investigative Site, Weiden
  - Novartis Investigative Site, Witten
  - Novartis Investigative Site, Wittenberg
- Greece (7):
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Voula, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chalcis
  - Novartis Investigative Site, Thessaloniki
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City
  - Novartis Investigative Site, Quetzaltenango
- Hong Kong (2):
  - Novartis Investigative Site, Pokfulam, Hong Kong
  - Novartis Investigative Site, Hong Kong
- Hungary (11):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Budapest, HUN
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Cegléd
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Makó
  - Novartis Investigative Site, Mátészalka
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Székesfehérvár
- Iceland (2):
  - Novartis Investigative Site, Kopavogur
  - Novartis Investigative Site, Reykjavik
- India (33):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Guntur, Andhrapradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Karamsad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Banglaore, Karnataka
  - Novartis Investigative Site, Bengaluru, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Kozhikode, Kerala
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Aurangabad, Maharashtra
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Wardha, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Dehradun, Uttarakhand
  - Novartis Investigative Site, Belagavi
  - Novartis Investigative Site, Coimbatore
  - Novartis Investigative Site, New Delhi
- Israel (6):
  - Novartis Investigative Site, Beersheba
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Giborim, Holon
- Italy (22):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Cinisello Balsamo, MI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
- Japan (16):
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Tsuchiura, Ibaraki
  - Novartis Investigative Site, Komatsu, Ishikawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Kawaguchi, Saitama
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
- Lebanon (4):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Hazmiyeh
  - Novartis Investigative Site, Saida
- Malaysia (3):
  - Novartis Investigative Site, Pulau Pinang, Pulau Pinang
  - Novartis Investigative Site, Kota Samarahan, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (8):
  - Novartis Investigative Site, Torreón, Coahulia
  - Novartis Investigative Site, Mexico City, Gustavo A Madero
  - Novartis Investigative Site, Cuernavaca, Morelos
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Distrito Federal
  - Novartis Investigative Site, Querétaro
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (16):
  - Novartis Investigative Site, Apeldoorn, DZ
  - Novartis Investigative Site, Sneek, The Netherlands
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Hardenberg
  - Novartis Investigative Site, Heemstede
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Venlo
- Norway (4):
  - Novartis Investigative Site, Moss
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Tynset
- Peru (12):
  - Novartis Investigative Site, Trujillo, La Libertad
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Chorrillos, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, Miraflores, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Juan de Miraflores, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
  - Novartis Investigative Site, Lima
  - Novartis Investigative Site, Piura
- Philippines (5):
  - Novartis Investigative Site, Davao City, Davao Region
  - Novartis Investigative Site, Cebu City
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
  - Novartis Investigative Site, San Juan City
- Poland (10):
  - Novartis Investigative Site, Warsaw, Masovian Voivodeship
  - Novartis Investigative Site, Elblag, Warmian-Masurian Voivodeship
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Kędzierzyn-Koźle
  - Novartis Investigative Site, Legnica
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Zabrze
- Portugal (4):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Covilha
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Setúbal
- Puerto Rico (2):
  - Novartis Investigative Site, Manatí
  - Novartis Investigative Site, Ponce
- Romania (14):
  - Novartis Investigative Site, Piteşti, Argeş
  - Novartis Investigative Site, Iași, Jud Iasi
  - Novartis Investigative Site, Târgu Mureş, Jud Mures
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Bacau
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Buzău
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Iași
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Târgu Mureş
- Russia (27):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Korolev Moscow Region
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Kursk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Pyatigorsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Sochy
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Troitsk Moscow Region
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Vladikavkaz
  - Novartis Investigative Site, Vsevolozhsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (32):
  - Novartis Investigative Site, Martin, Okr Martin
  - Novartis Investigative Site, Turčianske Teplice, Okr Turcianske Teplice
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Komárno, Slovak Republic
  - Novartis Investigative Site, Lučenec, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Rimavská Sobota, Slovak Republic
  - Novartis Investigative Site, Rožňava, Slovak Republic
  - Novartis Investigative Site, Svidník, Slovak Republic
  - Novartis Investigative Site, Handlová, SVK
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Brezno
  - Novartis Investigative Site, Dolný Kubín
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Piešťany
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Rimavská Sobota
  - Novartis Investigative Site, Sabinov
  - Novartis Investigative Site, Trebišov
  - Novartis Investigative Site, Trnava
  - Novartis Investigative Site, Žilina
  - Novartis Investigative Site, Žilina, Žilina Region
- Slovenia (3):
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Ljubljana
  - Novartis Investigative Site, Maribor
- South Africa (6):
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Lenasia, Gauteng
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Krugersdorp
- South Korea (11):
  - Novartis Investigative Site, Daegu, Dalseo Gu
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, KOR
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- Spain (17):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Cáceres, Extremadura
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Reus, Tarragona
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Huelva
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Sweden (4):
  - Novartis Investigative Site, Goethenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich
- Taiwan (7):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Hsinchu
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
  - Novartis Investigative Site, Yilan
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (10):
  - Novartis Investigative Site, Eskişehir, Meselik
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Haydarpasa Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Kucukcekmece/Istanbul
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Samsun
- United Kingdom (33):
  - Novartis Investigative Site, Peterborough, Cambridgeshire
  - Novartis Investigative Site, Stockton-on-Tees, Cleveland
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, Craigavon, Northern Ireland
  - Novartis Investigative Site, Axbridge, Somerset
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Chertsey, Surrey
  - Novartis Investigative Site, Sketty, Swansea
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Harrow
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Middlesex
  - Novartis Investigative Site, Milton Keynes
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Telford
  - Novartis Investigative Site, Tyne and Wear
  - Novartis Investigative Site, West Midlands
  - Novartis Investigative Site, Wiltshire
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No